CLINICAL TRIAL: NCT01154192
Title: Theca Cell Function in Adolescents With Polycystic Ovary Syndrome (PCOS)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: University of Virginia (Other)
Responsible Party: Principal Investigator, Jeffrey Chang, MD, Principal Investigator, University of California, San Diego
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 081696
Record Dates: First submitted 2010-06-29; First posted 2010-06-30 (Estimated); Results first posted 2019-04-23 (Actual); Last update posted 2019-04-30 (Actual); Status verified 2019-04

CONDITIONS: PCOS
Keywords: PCOS; oligomenorrhea; irregular menses; hyperandrogenemia; elevated testosterone; adolescents; androgens; ovary; LH
MeSH Terms: conditions — Oligomenorrhea; Menstruation Disturbances | interventions — Dexamethasone; Chorionic Gonadotropin; Ovidrel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- PCOS group (Experimental): Intervention: Each subject in the PCOS group will receive 1 mg of oral dexamethasone in the evening and return in the morning for an injection of 25ug of IV recombinant human chorionic gonadotropin. Subjects will also have blood drawn at times -0.5, 0, 0.5, and 24 hours after the injection of r-hCG for measurement of steroid hormones.
  Interventions: Drug: Dexamethasone; Drug: recombinant human chorionic gonadotropin (r-hCG)
- Normal group (Experimental): Intervention: Each subject in the Normal group will receive dexamethasone 1 mg orally in the evening and return the next morning for an injection of 25ug of IV recombinant human chorionic gonadotropin. Subjects will the have blood drawn at -0.5, 0, 0.5, and 24 hours after hCG injection for steroid hormone measurements.
  Interventions: Drug: Dexamethasone; Drug: recombinant human chorionic gonadotropin (r-hCG)
- Oligomenorrhea group (Experimental): Intervention: Each subject in the Oligomenorrhea group will receive dexamethasone 1 mg orally in the evening and return the next morning for an injection of 25ug of IV recombinant human chorionic gonadotropin. Subjects will the have blood drawn at -0.5, 0, 0.5, and 24 hours after hCG injection for steroid hormone measurements.
  Interventions: Drug: Dexamethasone; Drug: recombinant human chorionic gonadotropin (r-hCG)

INTERVENTIONS:
Drug: Dexamethasone — Each subject in each group will receive 1 mg of oral dexamethasone in the evening and return in the morning for an injection of 25ug of IV recombinant human chorionic gonadotropin. Subjects will also have blood drawn at times -0.5, 0, 0.5, and 24 hours after the injection of r-hCG for measurement of steroid hormones.
  Other Names: recombinant human chorionic gonadotropin (r-hCG)
Drug: recombinant human chorionic gonadotropin (r-hCG) — Each subject in each group will receive 1 mg of oral dexamethasone in the evening and return in the morning for an injection of 25ug of IV recombinant human chorionic gonadotropin (r-hCG). Subjects will also have blood drawn at times -0.5, 0, 0.5, and 24 hours after the injection of r-hCG for measurement of steroid hormones.
  Other Names: Ovidrel

SUMMARY:
In women with polycystic ovary syndrome (PCOS), the cardinal physiological abnormality is excessive ovarian androgen production marked by increased serum testosterone (T) and androstenedione (A) levels. Studies to determine the alteration in ovarian steroidogenesis that lead to abnormal production of ovarian androgens have revealed increased CYP17 gene expression with accentuated 17-hydroxylase activity leading to exaggerated 17-hydroxyprogesterone (17P) responses to luteinizing hormone (LH) stimulation. In contrast, T and A responses did not distinguish between PCOS and normal women, although these androgens were clearly greater in the former compared to the latter group. As a result, 17P responsiveness has been employed to determine the functional capacity of the ovary to produce androgens. The stimulatory agents that have been used included GnRH agonist, Lupron, at a dose of 10 microgram per kilogram, or hCG at a dose of 10,000 IU. The investigators propose to conduct a study that will determine the pattern of androgen responsiveness to 25ucg of hCG after 24 hours in adolescents with PCOS, those with oligomenorrhea, and in normal controls. This will allow for a comparison of these adolescents' ovarian functional capacity to produce androgens.

DETAILED DESCRIPTION:
In women with polycystic ovary syndrome (PCOS), the cardinal physiological abnormality is excessive ovarian androgen production marked by increased serum testosterone (T) and androstenedione (A) levels. Studies to determine the alteration in ovarian steroidogenesis that lead to abnormal production of ovarian androgens have revealed increased CYP17 gene expression with accentuated 17-hydroxylase activity leading to exaggerated 17-hydroxyprogesterone (17P) responses to luteinizing hormone (LH) stimulation. In contrast, T and A responses did not distinguish between PCOS and normal women, although these androgens were clearly greater in the former compared to the latter group. As a result, 17P responsiveness has been employed to determine the functional capacity of the ovary to produce androgens. The stimulatory agents that have been used included GnRH agonist, Lupron, at a dose of 10 microgram per kilogram, or hCG at a dose of 10,000 IU.We propose to conduct a study that will determine the pattern of androgen responsiveness to 25ucg of hCG after 24 hours in adolescents with PCOS, those with oligomenorrhea, and in normal controls. This will allow for a comparison of these adolescents' ovarian functional capacity to produce androgens.

ELIGIBILITY:
Inclusion Criteria:

* Normal CBC (Hemoglobin must be at least 11mg/dl)
* Normal renal and liver function tests
* Normal vital signs including normal blood pressure

Exclusion Criteria:

* Pregnancy
* On oral contraceptives
* On insulin lowering drugs
* On anti-androgens (i.e., spironolactone, flutamide, finasteride, etc)
* On medications that will influence androgen metabolism or clearance
* On medications that will inhibit the cytochrome P450 enzyme system (Cimetidine, ketoconazole, etc)

Ages: 12 Years to 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 24 (Actual)
Dates: Start 2011-08; Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R. Jeffery Chang, M.D., Principal Investigator — UCSD School of Medicine
Locations (1):
- UCSD School of Medicine, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- PCOS Group: Intervention: Each subject in the PCOS group will receive dexamethasone 1 mg orally in the evening and return the next morning for an injection of 25ug of IV recombinant human chorionic gonadotropin. Subjects will the have blood drawn at -0.5, 0, 0.5, and 24 hours after hCG injection for steroid hormone measurements.
  Dexamethasone: Each subject in each group will receive 1 mg of oral dexamethasone in the evening and return in the morning for an injection of 25ug of IV recombinant human chorionic gonadotropin. Subjects will also have blood drawn at times -0.5, 0, 0.5, and 24 hours after the injection of r-hCG for measurement of steroid hormones.
  recombinant human chorionic gonadotropin (r-hCG): Each subject in each group will receive 1 mg of oral dexamethasone in the evening and return in the morning for an injection of 25ug of IV recombinant human chorionic gonadotropin (r-hCG). Subjects will also have blood drawn at times -0.5, 0, 0.5, and 24 hours after the injection
- Normal Group: Intervention: Each subject in the Normal group will receive dexamethasone 1 mg orally in the evening and return the next morning for an injection of 25ug of IV recombinant human chorionic gonadotropin. Subjects will the have blood drawn at -0.5, 0, 0.5, and 24 hours after hCG injection for steroid hormone measurements.
  Dexamethasone
Period: Overall Study
Arm/Group | PCOS Group | Normal Group | There Were Only 2 Groups: PCOS and Normal Subjects
Started | 14 | 10 | 0
Completed | 14 | 10 | 0
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Oligpomenorrhea subjects not part of study
Groups:
- Total: Total of all reporting groups
Arm/Group | PCOS Group | Normal Group | Oligomenorrhea Group | Total
Number analyzed (Participants) | 14 | 10 | 0 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 14.9 (1.0) | 15.4 (1.2) |  | 15.3 (1.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 10 |  | 24
  Male | 0 | 0 |  | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: 17OHP Levels After hCG
Description: Assess serum levels of 17OHP after stimulation with recombinant hCG
Time Frame: 24 hours
Population: Oligmenorhea group not included in study
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | PCOS Group | Normal Group | Oligomenorrhea Group
Number analyzed (Participants) | 14 | 10 | 0
ng/ml | 3.2 (0.5) | 1.3 (0.3) |

2. Secondary Outcome: Testosterone
Description: Assess seruim levels of testosterone after stimulation with recombinant hCG
Time Frame: 24 hours
Population: Oligpmenrreha group not included in study
Measure: Mean (Standard Error); unit: ng/ml
Groups:
- Normal Group: Intervention: Each subject in the Normal group will receive dexamethasone 1 mg orally in the evening and return the next morning for an injection of 25ug of IV recombinant human chorionic gonadotropin. Subjects will the have blood drawn at -0.5, 0, 0.5, and 24 hours after hCG injection for steroid hormone measurements.
  .
Arm/Group | PCOS Group | Normal Group | Oligomenorrhea Group
Number analyzed (Participants) | 14 | 10 | 0
ng/ml | 1.6 (0.2) | 1.0 (0.2) |

3. Secondary Outcome: Androstenedione
Description: Assess serum levels of androstenedione after stimaultion with recombinant hCG
Time Frame: 24 hours
Population: Oligomenorreha group not inlcuded in study
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | PCOS Group | Normal Group | Oligomenorrhea Group
Number analyzed (Participants) | 14 | 10 | 0
ng/ml | 2.1 (0.2) | 0.9 (0.2) |

4. Secondary Outcome: DHEA
Description: Assess serum levels of DHEA after stimulation with recombinant hCG
Time Frame: 24 hours
Population: Oligomenrrhea group not included in study
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | PCOS Group | Normal Group | Oligomenorrhea Group
Number analyzed (Participants) | 14 | 10 | 0
ng/ml | 1.6 (0.2) | 1.0 (0.2) |

ADVERSE EVENTS:
Time Frame: 1 year
Description: The number of participants at risk for Other Adverse Events, All-Cause Mortality, and Serious Adverse Events should be 24
Groups:
- Oligomenorrhea Group: Not included in the study
Arm/Group | PCOS Group | Normal Group | Oligomenorrhea Group
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/10 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/10 | 0/0
Other Adverse Events (participants affected / at risk) | 0/14 | 0/10 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes